CLINICAL TRIAL: NCT02765997
Title: Single-Center, Open Label, Randomized Trial Comparing StemRegenin-1 Expanded Versus Unmanipulated Umbilical Cord Blood Transplantation In Patients With High-Risk Malignancy
Brief Title: StemRegenin-1 Expanded vs Unexpanded UCB for High Risk Heme Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Disapproval
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS006; MT2016-01 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelodysplasia
Keywords: AML; ALL; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unmanipulated UCB (Active Comparator): Subjects will receive unmanipulated umbilical cord blood transplantation after a myeloablative CY/FLU/TBI conditioning.
  Interventions: Biological: Unmanipulated UCB
- StemRegenin-1 UCB (Experimental): Subjects will receive StemRegenin-1 (SR-1) cultured umbilical cord blood transplantation after a myeloablative CY/FLU/TBI conditioning.
  Interventions: Biological: SR-1 UCB

INTERVENTIONS:
Biological: Unmanipulated UCB — Unmanipulated UCB infusion given on Day 0. All patients will receive the same conditioning and immunoprophylaxis for the prevention of acute and chronic GVHD, previously demonstrated to offer the best outcomes in recipients of partially HLA matched UCB. Standard supportive care, including the use of Neupogen [G-CSF] and prophylactic anti-bacterial, protozoal, viral and fungal agents, will also be prescribed. Supportive care will be modified throughout the transplant course at the treating physician's judgement.
  Other Names: Unmanipulated Umbilical Cord Blood
  Arms: Unmanipulated UCB
Biological: SR-1 UCB — SR-1 UCB infusion given on Day 0. All patients will receive the same conditioning and immunoprophylaxis for the prevention of acute and chronic GVHD, previously demonstrated to offer the best outcomes in recipients of partially HLA matched UCB. Standard supportive care, including the use of Neupogen [G-CSF] and prophylactic anti-bacterial, protozoal, viral and fungal agents, will also be prescribed. Supportive care will be modified throughout the transplant course at the treating physician's judgement.
  Other Names: StemRegenin-1 cultured umbilical cord blood
  Arms: StemRegenin-1 UCB

SUMMARY:
This is an open label, interventional, randomized phase II trial comparing StemRegenin-1 (SR-1) cultured umbilical cord blood (experimental arm) to unmanipulated umbilical cord blood (standard of care arm) transplantation after a myeloablative CY/FLU/TBI conditioning. A 2:1 randomization will be employed with a higher chance of being assigned to the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Must have a partially HLA matched UCB unit with a pre-cryopreserved TNC dose >2.5 x 107 per kilogram recipient weight. HLA matching is initially based on 4 of 6 HLA-A and B (at low or intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing).
* Eligible Diseases

  * Acute myelogenous leukemia (AML) at the following stages:

    * Intermediate to high risk leukemia in first complete remission (CR1) based on institutional criteria.
    * Any second or subsequent CR.
    * Secondary AML with prior malignancy that has been in remission for at least 12 months.
  * Acute lymphocytic leukemia (ALL) at the following stages:

    * High risk first remission.

      1. Ph+ ALL, or
      2. MLL rearrangement with slow early response at Day 14, or
      3. Hypodiploidy (< 44 chromosomes or DNA index < 0.81), or
      4. End of induction M3 bone marrow, or
      5. End of induction M2 with M2-3 at Day 42.
    * High risk second CR based on institutional criteria (eg, for children, bone marrow relapse <36 months from induction or T-lineage bone marrow relapse or very early isolated central nervous system (CNS) relapse <6 months from diagnosis, or slow re-induction (stage M2-3 at day 28 after induction) regardless of length remission.
    * Any third or subsequent CR.
  * Biphenotypic/undifferentiated leukemia in CR
  * Chronic myelogenous leukemia (CML) excluding refractory blast crisis
  * Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt) or refractory anemia
* Other Inclusion Criteria

  * Karnofsky score >70% (16 years and older) or a Lansky play score >70 (children <16 years) - appendix II
  * Adequate organ function defined as:

    * Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) >70 mL/min/1.73 m2.
    * Hepatic: Bilirubin ≤2.5 x mg/dL; AST, ALT, alkaline phosphatase <5 x upper limit of normal,
    * Pulmonary function: DLCO, FEV1, FEC (diffusion capacity) >50% of predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then normal O2 saturation on room air.
    * Cardiac: Left ventricular ejection fraction at rest must be >45%
  * Available 'back-up' HSPC graft (e.g, second partially HLA matched UCB unit, haploidentical related donor).
  * Voluntary written consent signed (adult or parental) before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Females of childbearing potential must have a blood test or urine study within 14 days prior to study enrollment to rule out pregnancy.
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology.
* Active bacterial, viral or fungal infection (currently taking medication and progression of clinical symptoms).
* Prior autologous or allogeneic transplant within past 12 months.
* Other active malignancy.
* Inability to receive TBI 1320 cGy (e.g., extensive prior therapy including >12 months alkylator therapy or >6 months alkylator therapy with extensive radiation. Or prior Y-90 ibritumomab (Zevalin) or I-131 tostumomab (Bexxar), as part of their salvage therapy.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Recovery | Day 14 after transplantation
  Percentage of patients with neutrophil recovery

SECONDARY OUTCOMES:
Secondary Graft Failure | Day 100 after transplantation
  Percentage of patients with secondary graft failure
Platelet Recovery | Day 100 after transplantation
  Percentage of patients with platelet recovery
Transplant-Related Mortality | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: John Wagner, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States